CLINICAL TRIAL: NCT06489561
Title: Probing the Neural Computations Underlying Goal-directed Decision-making in Humans With Single-neuron Recordings
Brief Title: Neural Computations of Goal-directed Decision-making
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); California Institute of Technology (Other)
Responsible Party: Principal Investigator, Adam Mamelak, MD, Staff Physician III, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MOD00001351; R01MH133729 (NIH)
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy Intractable
Keywords: Epilepsy; Decision-making; Depth Electrode
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioral Testing (Experimental): Behavioral and Neuronal Recordings
  Interventions: Behavioral: Cedrus RB-844 response pad; Adtech Behnke-Fried micro-electrodes; Neurolynx electrophysiology system

INTERVENTIONS:
Behavioral: Cedrus RB-844 response pad; Adtech Behnke-Fried micro-electrodes; Neurolynx electrophysiology system — Devices listed are components of a single intervention that includes: Record patient responses (Cedrus RB-844), record neuronal activity (Neurolynx) from electrodes (Adtech Behnke-Fried)

SUMMARY:
The purpose of this research is to better understand how the human brain accomplishes the cognitive task of making goal-directed decisions. These investigations are critical to better understand human cognition and to design treatments for disorders of decision making and performance monitoring.

DETAILED DESCRIPTION:
Flexible goal-directed decision-making is a core aspect of higher-order adaptive biological intelligence. A number of psychiatric disorders involve impairments in goal-directed decision-making, yet the current lack of even a basic understanding of how goal-directed action selection is implemented at the neuronal level in humans hinders the ability to pinpoint these neuropsychiatric dysfunctions. In particular, it is completely unknown how goals, and the stimuli and actions that need to be selected from in order to pursue them, are represented at the level of single neurons, nor how goals get selected from available possible goals.

The study experiments utilize the rare opportunity to record in-vivo from human single neurons simultaneously in multiple brain areas in patients undergoing treatment for drug resistant epilepsy. The study will utilize a combination of (i) in-vivo recordings in awake behaving humans assessing decision making accuracy and ability through choice ratings, (ii) computational analysis and modeling.

These techniques will be applied to characterize the functional contribution of human ventromedial prefrontal (vmPFC), dorsal anterior cingulate (dACC) and pre-supplementary motor area (pre-SMA) in these processes. Investigators will first test the longstanding proposal never tested at the neuronal level in humans that the value of stimuli is especially represented by neurons in vmPFC, while the value of actions are more represented by neurons in dorsal cortical areas such as the pre-SMA. Investigators will then address how goals themselves are represented. In the real world, animals including humans need to select a goal before any action is performed. Thus, there is a hierarchical process of goal selection followed by action selection. Investigators hypothesize that the vmPFC plays a specific role in goal-valuation and selection, while neurons in dorsomedial areas including pre-SMA and dACC will play more of a role in valuing and selecting the actions that implement the chosen goal.

The expected outcome of this work is a comprehensive understanding of the functions of the human PFC in goal-directed decision-making at cellular resolution while shedding light on the neural mechanisms of goal-representation and selection which hitherto has been virtually unstudied.

ELIGIBILITY:
Inclusion Criteria:

* Intractable epilepsy, undergoing invasive monitoring
* Age ≥13
* Full Scale Intelligence Quotient > 70
* Ability to comprehend and perform simple behavioral tasks by pressing buttons on laptop computer in response to questions

Exclusion Criteria:

* Determination by clinicians and investigators that a patient is unable to complete the behavioral tasks required for the protocol due to either cognitive limits, psychological limits, or pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Decision Making (Firing Rates) | 5 years
  Neuronal firing rates of cells (measured in spike rates per second) in the frontal lobes during a decision-making process.
Decision Making (Power) | 5 years
  Power of local field potential bandwidths (measured in amplitude across frequency of the bandwidths) in the frontal lobes during a decision-making process.
Decision Making (Timing) | 5 years
  Timing of neuronal discharges (measured in spike rates per second) across the frontal lobes during a decision-making process.

CONTACTS AND LOCATIONS:
Overall Officials: Ueli Rutishauser, PhD, Principal Investigator — Cedars-Sinai Medical Center; Adam Mamelak, MD, Principal Investigator — Cedars-Sinai Medical Center; John O'Doherty, PhD, Principal Investigator — California Institute of Technology
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No